CLINICAL TRIAL: NCT02631616
Title: Treatment With Sandostatin in Patients With Castrate Resistance Prostate Cancer Showing Uptake of 68Ga-DOTATET
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ofer Gofrit, Prof. Ofer N. Gofrit, MD, PhD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPros-HMO-CTIL
Record Dates: First submitted 2015-12-03; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasma, Castration-Resistant; neuroendocrine differentiation; 68Ga-DOTATET; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): Monthly injections of Somatostatin (Sandoatatin LAR - 30mg)
  Interventions: Drug: Somatostatin

INTERVENTIONS:
Drug: Somatostatin — Monthly injections of Somatostatin
  Other Names: Sandoatatin LAR - 30mg

SUMMARY:
Purpose: Castrate resistance prostate cancer (CRPC) often shows histological evidence of neuroendocrine differentiation (NED). Recently the investigators initiated a research project investigating the uptake of the radiotracer 68Ga-DOTATET (a marker of neuroendocrine tumors-NET) in PET/CT in patients with CRPC. In 4/8 patients studied thus far, uptake of the tracer in bone metastases was found. It has been shown that monthly injections of Somatostatin lengthen overall survival in patients with NET. The purpose of the current project is to examine the ability of Somatostatin to stabilize or possibly reverse metastases in patients with CRPC that express high level of somatostatin receptors in 68Ga-DOTATET PET/CT.

Materials and Methods: 30 patients with CRPC will be studied with 68Ga-DOTATET PET/CT. Patients showing uptake of the radiotracer 68Ga-DOTATET in at two least to metastases will be considered eligible for the study. These patients will be evaluated biochemically and clinically and will be treated with monthly injections of Sandoatatin LAR - 30mg. Clinical, biochemical and imaging studies (68Ga-DOTATET PET/CT) will be repeated after 4 and 12 months of treatment. Responding patients (stabilization or decrease in the number and SUV of metastases) will be subjected to continued therapy until progression.

DETAILED DESCRIPTION:
Introduction: Neuroendocrine tumors (NET) present receptors to somatostatin. This feature is utilized therapeutically in patients with metastatic NET. Monthly injection of Somatostatin was shown to lengthen overall survival (compared to placebo) in these patients. From histological studies it is known that advanced prostate cancer often shows neuroendocrine differentiation (NED). This is considered one of the mechanisms of "escape" of tumor cells from androgen deprivation therapy. Recently the investigatros initiated a research project investigating the uptake of the radiotracer 68Ga-DOTATET (a marker of neuroendocrine tumors-NET) in PET/CT in patients with castrate resistance prostate cancer. In 4/8 patients studied thus far, uptake of the tracer in bone metastases was found.

Purpose: The purpose of the current project is to examine the ability of LAR Somatostatin to stabilize or possibly reverse metastases in patients with castrate resistance prostate cancer that express high level of somatostatin receptors.

The aims of the study are:

1. To detect biochemical response (PSA and chromogranin A)
2. To detect PET response (in repeated PET/CT, 68Ga-DOTATET).
3. To detect clinical response (QOL 30 questioner).
4. To detect adverse response.

Materials and Methods:

1. Eligible patients will be evaluated by: serum levels of PSA, chromogranin A, Pro GRP and possibly other non-genetic markers and by QOL 30 questioner
2. Treatment with monthly injections of Sandoatatin LAR - 30mg will be initiated.
3. Evaluation will be done after 4 injections and will include: blood tests for PSA and chromogranin A, Pro GRP and possibly other non-genetic markers and by QOL 30 questioner and by PET/CT with 68Ga-DOTATET. Similar evaluation will be done after 12 injections. Responding patients (stabilization or decrease in the number and SUV of metastases) will be subjected to continued therapy until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven prostate cancer.
2. Hormonal treatment (either surgical orchiectomy or medical castration with LHRH agonist or antagonist).
3. Proven castration levels (serum Testosterone< 50 ng/dl)
4. Radiological evidence of metastatic disease.
5. Uptake of the radiotracer 68Ga-DOTATET in at two least to metastases.

Exclusion Criteria:

1. Participation in another trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 4 months
  QOL 30 questioner

SECONDARY OUTCOMES:
Biochemical response | 4 months
  Blood test for PSA (in ng/ml)
Imaging response | 4 months
  PET/CT with 68Ga-DOTATET

IPD SHARING:
Plan to Share IPD: Undecided